CLINICAL TRIAL: NCT06283199
Title: The Importance of Ecological Momentary Assessment to Capture the Whole Patient's Symptoms Experience in Musculo-skeletal Conditions
Brief Title: Comparing Reports Recorded by the Patients at the Time at Which They Feels Pain to What Patients Report at Monthly Visits to Assess Symptoms of Musculoskeletal Diseases.
Status: Recruiting | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Other Study IDs: ORL-ORT-025
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients will be introduced to the use of a mobile application for their smartphone to record the Ecological Momentary Assessment (EMA). This app will ask the patients to assess their pain and function two times daily for 2 months.

After 1 month and at the end of the 2 months, follow-up visits will be performed and patients will be asked to retrospectively evaluate the pain that they suffered and the level of function they had during the last month.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients
* Patients able to give informed consent and to follow the protocol of the study (i.e. able to use a smartphone)
* Patients >18 years
* BMI <35 and >18.5
* Patients with a smartphone with Android or iOS as operative systems

Exclusion Criteria:

* Patients unable to follow the protocol of the study (i.e. unable to use a smartphone, not owning a smartphone or unwilling to download or use the application)
* Patients with a diagnosis of a musculoskeletal injury but without symptoms
* Patients without a radiological examination confirming the diagnosis of musculoskeletal disease
* Patients with planned surgery in the following 60 days
* Pregnant or lactating woman
* Patients with other diseases causing pain in the involved joint (e.g. rheumatoid arthritis or other rheumatologic diseases).
* Surgical treatment in the last year and intra-articular injection in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with musculoskeletal chronic pain with a clinical and imaging diagnosis of an orthopaedic disease such as knee osteoarthritis, hip osteoarthritis, shoulder osteoarthritis, ankle osteoarthritis, rizoathrosis, meniscectomy treatment, rotator cuff tendinopathy, low-back pain, Achille tendinopathy, patellar tendinopathy,and tennis elbow.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in pain level | one month
  difference between the level of pain collected within the first month of mobile application and the level of pain reported through a retrospective recall-based assessment on the 0-10 Numerical Rating Scale

CONTACTS AND LOCATIONS:
Locations (2):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy
- EOC - Orthopaedics and Traumatology Service, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No